CLINICAL TRIAL: NCT04453527
Title: The CASCADE Study - Measures of Complement Activation and Inflammation in Patients With Coronavirus Disease 2019
Brief Title: The CASCADE Study - Measures of Complement Activation and Inflammation in Patients With Covid-19
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Akari Therapuetics (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/37
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is a new disease and therefore it is still not clear exactly how the virus affects the body and why people are affected so differently. It causes infection in the lungs and the virus can then attack blood vessels in the lungs and other organs to spark off an inflammatory process that can make a person very ill. It also can cause damage within tiny blood vessels that makes a person's blood thicken up and stop flow in vital organs. The investigators believe complement (which is a chemical in the body which can be harmful in excess) orchestrates the inflammation and thickening of the blood that can make a person sick. The investigators now need to know which of these complement chemicals are elevated in COVID-19 and compare to healthy volunteers, and assess whether the levels are higher in people with severe lung disease. The investigators believe that if levels are increased there are special treatments that can counteract them and potentially be an effective treatment for COVID-19.

In this study the investigators will measure different parts of the inflammation process to better understand what may be causing severe disease and to see if there may be benefits from a new treatment to reduce inflammation

DETAILED DESCRIPTION:
This study is an observational cross-sectional and cohort study to assess whether there is evidence of increased complement activation and/or LTB4 levels and other parameters of inflammation and a pro-coagulative state in adult patients hospitalised with COVID-19 compared to healthy controls and also whether these measures differ with increasing severity of respiratory failure.

Blood samples (serum and plasma) will be obtained from each participant at the time of recruitment into the trial, to assess the profile of complement activation, cytokines/ chemokines, leukotrienes (specifically leukotriene B4) and markers of coagulation and inflammation in patients with COVID-19.

Participants within the cohort study will be recruited at the point of admission or as close to it as possible. Baseline sampling will be performed at time of recruitment. There will be up to 2 additional sampling points (with not more than one sample per day) if there is any worsening of the participants respiratory failure (i.e. deteriorating from mild to moderate or moderate to severe disease).

Patients just admitted to hospital will be asked to consent for both the case control and the cohort study

Data will be collected at baseline for all participants and then again at each further sampling point for the participants within the cohort study.

Patient status will be measured at 14 days from the last point of sampling.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adults ≥18 years old requiring hospital admission for COVID-19

2. COVID-19 confirmed by either*:

* A positive swab (using RT-PCR)
* OR based on a high level of clinical probability confirmed by the presence of typical symptoms and compatible radiological findings on imaging with no alternative cause for these findings identified by the treating physician.

Exclusion Criteria:

* 1. Renal replacement therapy on ITU

  2. Significant trauma (including an acute fracture or significant head injury)

  3. Massive transfusion of blood products

  4. Confirmed bacteraemia with pathogenic organism on blood cultures or other severe bacterial infections (including abscess/empyema) which persist despite broad-spectrum antibiotics and are thought to be significantly contributing to the patient's symptoms and clinical state. Recruitment will not be delayed however pending a negative culture.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with Covid 19 and Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Complement Activation | 14 days sampling time period
  C5a, C5, C3, sC5b9, Bb concentration from serum
Leukotrienes Measure | 14 days sampling time period
  LTB4 concentration from plasma
Coagulation Measure | 14 days sampling time period
  Level of platelets, INR, APTS, D-Dimer, Fibrinogen, thrombin antithrombin complex (TAT), from citrate plasma
Hyperinflammation Measure | 14 days sampling time period
  • CRP, Ferritin, PCT, LDH, Troponin, ALT from plasma
Cell Count | 14 days sampling time period
  Total White Blood Cell count (including lymphocytes, monocytes and neutrophils)
Cytokines and Chemokine Measure | 14 days sampling time period
  Level of • Pro-inflammatory - IL-1α, IL-1β, IL-2, IL-5, IL-6, IL-7, IL-8, IL-17, GCSF, GMCSF, IFN γ, IP10, MCP-1, MIP1α, TNFα and anti inflammatory IL-4, IL-10, IL-13, IL-22, TGF-α from plasma
Endothelial dysfunction measures: | 14 days sampling time period
  VEGF, tissue factor and PAI-1, from plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiffen L, D'Cruz LG, Brown T, Higenbottam TW, Bernstein JA, Campbell C, Moellman J, Ghosh D, Richardson C, Weston-Davies W, Chauhan AJ. Clinical severity classes in COVID-19 pneumonia have distinct immunological profiles, facilitating risk stratification by machine learning. Front Immunol. 2023 Sep 5;14:1192765. doi: 10.3389/fimmu.2023.1192765. eCollection 2023. PMID 37731491